CLINICAL TRIAL: NCT06559865
Title: Impact of a Paced Breathing Exercise Intervention on Autonomic Nervous System Function and Symptom Severity in Youth Post-concussion: a Pilot Feasibility Study
Brief Title: Impact of a Paced Breathing Exercise Intervention on Autonomic Nervous System Function After Pediatric Concussion
Acronym: Breathe
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Isabelle Gagnon, Senior Scientist, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-10503
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Concussion, Mild
MeSH Terms: conditions — Brain Concussion | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Breathing exercises (Experimental): In addition to the standard rehabilitation care in the concussion clinic, the intervention group will have a daily 10-minutes paced breathing home-exercise program. The paced breathing exercise including inhale for 4-second and exhale for 6-seconds, for a total of 6 breaths per minute.
  Interventions: Behavioral: Breathing exercises
- Usual care (No Intervention): Treatment for a concussion involves relative physical and cognitive rest for 24-48 hs, then a focus on gradually returning to normal activities and school as symptoms improve. Follow-up with healthcare professionals in the concussion clinic to ensure a safe and effective recovery and full return to school and sport. The concussion clinic follow-up includes meeting with a coordinator and physical therapist, and with a psychologist or MD if necessary

INTERVENTIONS:
Behavioral: Breathing exercises — as per group description
  Arms: Breathing exercises

SUMMARY:
The goal of this pilot clinical trial is to assess the feasibility of administering a paced breathing exercise intervention program to children and adolescents in the sub-acute period after concussion, and to document the autonomic function, and symptom severity (post-concussion symptoms, anxiety, sleep) before and after administration of the intervention.

Participants will:

will be instructed to perform a daily 10-minutes daily paced breathing home-exercise program and to document the daily exercises performed within a performance log, or receive usual care from a concussion follow-up program.

A weekly phone meeting will be performed with the participants, to review exercise, providing, specific instructions, and making any necessary adjustments.

All participants (intervention and control group) will undergo a second assessment after four weeks following completion of the intervention program. During the second assessment information regarding the intervention feasibility, time to return to school, return to sport, and clear from medication will be collected as well.

ELIGIBILITY:
Inclusion Criteria:

* aged 9-18 years
* seven days-3 months post-concussion,
* at least one post-concussion symptom in the Post-concussion Symptom Inventory (PSCI) that is relevant to ANS dysfunction (e.g. dizziness, nausea, fatigue, confusion, anxiety or sleep disturbances).

Exclusion Criteria:

* known heart disease,
* previous neurological problems other than concussion

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Feasibility-days of practice | 4 weeks
  number of days children in the experimental group will engage in performing their breathing exercises
Feasibility-daily duration of practice | 4 weeks
  number of minutes children in the experimental group will engage in performing their breathing exercises

SECONDARY OUTCOMES:
Autonomic nervous system function-Heart rate | initial and 4 week evaluation
  heart rate during autonomous nervous system testing
Autonomic nervous system function-Heart rate variability | initial and 4 week evaluation
  heart rate variability during autonomous nervous system testing

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University Health Center, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No